CLINICAL TRIAL: NCT03189342
Title: Effects of Dual-Task Training and Exercise-Cognitive Activity Combined Training on Fall Risk and Balance Performance in Elderly at Risk of Falls: A Randomised Controlled Trial Study
Brief Title: Effects of Training on Fall Risk and Balance Performances
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, leyla atas balci, Principal Investigator, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: E.4629
Record Dates: First submitted 2017-06-14; First posted 2017-06-16 (Actual); Last update posted 2017-06-16 (Actual); Status verified 2017-06

CONDITIONS: Accidental Falls
Keywords: Balance; Dual-task interference; Falls; Gait; Older Adults

STUDY DESIGN:
Intervention Model Description: Exercise training The volunteers were assigned to one of three interventions for 4 weeks. Group 1 performed balance and gait exercises. Group 2 performed cognitive activity simultaneously with balance and gait exercises. Group 3 performed cognitive, balance and gait activity training asynchronously at different times during the same day.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Single Task Training (Experimental): Performed balance and gait exercises
  Interventions: Behavioral: Single task training
- Dual task training (Experimental): Performed cognitive activity simultaneously with balance and gait exercises
  Interventions: Behavioral: dual task training
- Exercise-Cognitive Activity Combined Training (Experimental): Performed cognitive, balance and gait activity training asynchronously at different times during the same day
  Interventions: Behavioral: exercise-cognitive activity combined training

INTERVENTIONS:
Behavioral: Single task training — The participants in single task training received 30 minutes single task balance and gait exercises, 3 times a week for 4 weeks. The program included static and dynamic balance exercises. Static balance exercises involved body stability (e.g., standing legs open and closed, standing with eyes closed, tandem standing, standing on foam surface and one leg standing, standing while throwing and catching a ball ), forward and backward weight shifting and keeping standing position while being disturbed by external perturbation. Dynamic balance exercises included tandem walking, walking to different direction (backward, side to side), transfer activities (from 1 chair to another) and sit to stand 5 times
  Arms: Single Task Training
Behavioral: dual task training — The participants practiced 30 minutes balance and gait exercises while simultaneously performing cognitive tasks. The program included static and dynamic balance exercises. Static balance exercises involved body stability, forward and backward weight shifting and keeping standing position while being disturbed by external perturbation. Dynamic balance exercises included tandem walking, walking to different direction, transfer activities and sit to stand 5 times. The participants practiced cognitive tasks while simultaneously performing balance and gait exercises. The cognitive tasks included visual attention, auditory attention, planning, verbal fluency, simple mental math and maze activities. At each week, participants performed different type of activities which were designed to foster the executive functions: (1) Visual and auditory attention, (2) Planning and verbal fluency, (3) Simple math problems (4) Visual and auditory attention, planning, verbal fluency, math problems
  Arms: Dual task training
Behavioral: exercise-cognitive activity combined training — The participants first practiced 30 min of cognitive activities then performed 30 min of balance and gait exercises after 5 min of resting.The program included static and dynamic balance exercises. Static balance exercises involved body stability, forward and backward weight shifting and keeping standing position while being disturbed by external perturbation. Dynamic balance exercises included tandem walking, walking to different direction, transfer activities and sit to stand 5 times. The cognitive tasks included visual attention, auditory attention, planning, verbal fluency, simple mental math and maze activities. At each week, participants performed different type of activities which were designed to foster the executive functions: (1) Visual and auditory attention, (2) Planning and verbal fluency, (3) Simple math problems (4) Visual and auditory attention, planning, verbal fluency, math problems.
  Arms: Exercise-Cognitive Activity Combined Training

SUMMARY:
Dual task training has been shown to reduce the risk of falls more than single task training. However, there have been no studies which compared the effects of single task training, dual task training and asynchronous cognitive, balance exercise training during same day on the risk of falls among healthy older individuals. Therefore, the aim of this study was to investigate differences among the effects of single task training, dual task training and exercise-cognitive activity combined training on balance and gait performances and fall risk in elderly at risk of fall.

DETAILED DESCRIPTION:
The term "dual task" refers to the ability of performing 2 tasks simultaneously, for example, a cognitive and a motor task. Previous studies demonstrated that dual task training is more effective than single task training in reducing falls among elderly. These studies demonstrated that the improvements in balance and gait speed resulted in a decrease of fall frequency. Although dual task training has been shown to reduce the risk of falls more than single task training, to date, there have been no studies which compared the effects of single task training, dual task training and asynchronous cognitive, balance exercise training during same day on the risk of falls among healthy older individuals. Therefore, the aim of this study was to investigate differences among the effects of single task training, dual task training and exercise-cognitive activity combined training on balance and gait performances and fall risk in elderly at risk of fall.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 years or older
* literate
* having a fall incident during the past year
* ability to walk 10 meter without any support
* getting more than 13.5 seconds at Timed up and Go test
* getting less than 24 points at Standardized Mini-Mental State Examination

Exclusion Criteria:

* neurological or musculoskeletal diagnosis such as Parkinson's or Alzheimer's disease,
* orthopaedic involvement or significant visual and auditory impairments

Ages: 65 Years to 83 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 45 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Gait speed under single task condition | 4 weeks
  The participants walked 10 meter at their comfortable speed and the time to complete the task was recorded
Gait speed under dual task condition | 4 weeks
  The participants walked 10 meter while producing words which started with letter "K"
Timed Up and Go test | 4 weeks
  Timed Up and Go Test is a simple test used to measure mobility. The time required to stand up from a chair, walk 3 m to the line on the floor at a normal pace, walk back to the chair and sit down is measured (Thrane et al 2007)
Berg Balance Scale | 4 weeks
  The Berg Balance Scale (BBS) consists of 14 simple balance related tasks that measure the static, dynamic, and functional balance skills (Sahin et al 2008)
Falls Efficacy Scale | 4 weeks
  Tinetti's Falls Efficacy Scale (FES), which was used to assess fall-related self-efficacy, is a 10-questions scale (Scheffer et al 2008).

CONTACTS AND LOCATIONS:
Locations (1):
- Medipol Mega University Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is no plan to share data for other researches

REFERENCES:
- [Background] WHO Global Report on Falls Prevention in Older Age. 2007. Geneva, Switzerland: World Health Organization
- [Background] Falls, Fact sheet N°344. October 2012. World Health Organization
- [Background] What are the main risk factors for falls amongst older people and what are the most effective interventions to prevent these falls. 2004. Geneva, Switzerland: World Health Organization
- [Background] Rubenstein LZ. Falls in older people: epidemiology, risk factors and strategies for prevention. Age Ageing. 2006 Sep;35 Suppl 2:ii37-ii41. doi: 10.1093/ageing/afl084. PMID 16926202
- [Background] Austin N, Devine A, Dick I, Prince R, Bruce D. Fear of falling in older women: a longitudinal study of incidence, persistence, and predictors. J Am Geriatr Soc. 2007 Oct;55(10):1598-603. doi: 10.1111/j.1532-5415.2007.01317.x. PMID 17908062
- [Background] Tinetti ME, Kumar C. The patient who falls: "It's always a trade-off". JAMA. 2010 Jan 20;303(3):258-66. doi: 10.1001/jama.2009.2024. PMID 20085954
- [Background] Karlsson MK, Vonschewelov T, Karlsson C, Coster M, Rosengen BE. Prevention of falls in the elderly: a review. Scand J Public Health. 2013 Jul;41(5):442-54. doi: 10.1177/1403494813483215. Epub 2013 Apr 3. PMID 23554390
- [Background] Hardy SE, Perera S, Roumani YF, Chandler JM, Studenski SA. Improvement in usual gait speed predicts better survival in older adults. J Am Geriatr Soc. 2007 Nov;55(11):1727-34. doi: 10.1111/j.1532-5415.2007.01413.x. Epub 2007 Oct 3. PMID 17916121
- [Background] Guedes RC, Dias RC, Pereira LS, Silva SL, Lustosa LP, Dias JM. Influence of dual task and frailty on gait parameters of older community-dwelling individuals. Braz J Phys Ther. 2014 Sep-Oct;18(5):445-52. doi: 10.1590/bjpt-rbf.2014.0034. Epub 2014 Sep 12. PMID 25372007
- [Background] Chang JT, Morton SC, Rubenstein LZ, Mojica WA, Maglione M, Suttorp MJ, Roth EA, Shekelle PG. Interventions for the prevention of falls in older adults: systematic review and meta-analysis of randomised clinical trials. BMJ. 2004 Mar 20;328(7441):680. doi: 10.1136/bmj.328.7441.680. PMID 15031239
- [Background] Plummer P, Zukowski LA, Giuliani C, Hall AM, Zurakowski D. Effects of Physical Exercise Interventions on Gait-Related Dual-Task Interference in Older Adults: A Systematic Review and Meta-Analysis. Gerontology. 2015;62(1):94-117. doi: 10.1159/000371577. Epub 2015 Feb 19. PMID 25721432
- [Background] Wang X, Pi Y, Chen P, Liu Y, Wang R, Chan C. Cognitive motor interference for preventing falls in older adults: a systematic review and meta-analysis of randomised controlled trials. Age Ageing. 2015 Mar;44(2):205-12. doi: 10.1093/ageing/afu175. Epub 2014 Nov 5. PMID 25377745
- [Background] Thrane G, Joakimsen RM, Thornquist E. The association between timed up and go test and history of falls: the Tromso study. BMC Geriatr. 2007 Jan 12;7:1. doi: 10.1186/1471-2318-7-1. PMID 17222340
- [Background] Keskinoğlu P, Uçku R and Yener G. Pretest Results of the Revised Standardized Mini Mental Examination Test in Community Dwelling Elderly. Journal of Neurological Sciences 2008; 25: 18-24
- [Background] Shubert TE, Schrodt LA, Mercer VS, Busby-Whitehead J, Giuliani CA. Are scores on balance screening tests associated with mobility in older adults? J Geriatr Phys Ther. 2006;29(1):35-9. PMID 16630375
- [Background] Scheffer AC, Schuurmans MJ, van Dijk N, van der Hooft T, de Rooij SE. Fear of falling: measurement strategy, prevalence, risk factors and consequences among older persons. Age Ageing. 2008 Jan;37(1):19-24. doi: 10.1093/ageing/afm169. PMID 18194967
- [Background] Sahin F, Yilmaz F, Ozmaden A, Kotevolu N, Sahin T, Kuran B. Reliability and validity of the Turkish version of the Berg Balance Scale. J Geriatr Phys Ther. 2008;31(1):32-7. doi: 10.1519/00139143-200831010-00006. PMID 18489806
- [Background] Silsupadol P, Shumway-Cook A, Lugade V, van Donkelaar P, Chou LS, Mayr U, Woollacott MH. Effects of single-task versus dual-task training on balance performance in older adults: a double-blind, randomized controlled trial. Arch Phys Med Rehabil. 2009 Mar;90(3):381-7. doi: 10.1016/j.apmr.2008.09.559. PMID 19254600
- [Background] Silsupadol P, Siu KC, Shumway-Cook A, Woollacott MH. Training of balance under single- and dual-task conditions in older adults with balance impairment. Phys Ther. 2006 Feb;86(2):269-81. PMID 16445340
- [Background] Shumway-Cook A, Baldwin M, Polissar NL, Gruber W. Predicting the probability for falls in community-dwelling older adults. Phys Ther. 1997 Aug;77(8):812-9. doi: 10.1093/ptj/77.8.812. PMID 9256869
- [Background] Shumway-Cook A, Brauer S, Woollacott M. Predicting the probability for falls in community-dwelling older adults using the Timed Up & Go Test. Phys Ther. 2000 Sep;80(9):896-903. PMID 10960937
- [Background] Patil R, Uusi-Rasi K, Kannus P, Karinkanta S, Sievanen H. Concern about falling in older women with a history of falls: associations with health, functional ability, physical activity and quality of life. Gerontology. 2014;60(1):22-30. doi: 10.1159/000354335. Epub 2013 Oct 8. PMID 24107382
- [Background] Halvarsson A, Oddsson L, Olsson E, Faren E, Pettersson A, Stahle A. Effects of new, individually adjusted, progressive balance group training for elderly people with fear of falling and tend to fall: a randomized controlled trial. Clin Rehabil. 2011 Nov;25(11):1021-31. doi: 10.1177/0269215511411937. Epub 2011 Aug 17. PMID 21849377
- [Background] Halvarsson A, Franzen E, Stahle A. Balance training with multi-task exercises improves fall-related self-efficacy, gait, balance performance and physical function in older adults with osteoporosis: a randomized controlled trial. Clin Rehabil. 2015 Apr;29(4):365-75. doi: 10.1177/0269215514544983. Epub 2014 Aug 20. PMID 25142277
- [Background] Ruthruff E, Van Selst M, Johnston JC, Remington R. How does practice reduce dual-task interference: integration, automatization, or just stage-shortening? Psychol Res. 2006 Mar;70(2):125-42. doi: 10.1007/s00426-004-0192-7. Epub 2004 Nov 17. PMID 16703392
- [Background] Sherrington C, Whitney JC, Lord SR, Herbert RD, Cumming RG, Close JC. Effective exercise for the prevention of falls: a systematic review and meta-analysis. J Am Geriatr Soc. 2008 Dec;56(12):2234-43. doi: 10.1111/j.1532-5415.2008.02014.x. PMID 19093923
- [Background] van het Reve E, de Bruin ED. Strength-balance supplemented with computerized cognitive training to improve dual task gait and divided attention in older adults: a multicenter randomized-controlled trial. BMC Geriatr. 2014 Dec 15;14:134. doi: 10.1186/1471-2318-14-134. PMID 25511081
- [Background] Voelcker-Rehage C, Alberts JL. Effect of motor practice on dual-task performance in older adults. J Gerontol B Psychol Sci Soc Sci. 2007 May;62(3):P141-8. doi: 10.1093/geronb/62.3.p141. PMID 17507581
- [Derived] Drahota A, Udell JE, Mackenzie H, Pugh MT. Psychological and educational interventions for preventing falls in older people living in the community. Cochrane Database Syst Rev. 2024 Oct 3;10(10):CD013480. doi: 10.1002/14651858.CD013480.pub2. PMID 39360568